CLINICAL TRIAL: NCT04712045
Title: Rational Use of Personal Protective Equipment: a Randomised Trial and Quality Improvement Intervention During COVID-19 Pandemic
Brief Title: Rational Use of Personal Protective Equipment During COVID-19 Pandemic
Acronym: RUPERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, ProfessorPeterMcculloch, Professor of Surgical Science and Practice, University of Oxford
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRAS287865
Record Dates: First submitted 2021-01-11; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Personal Protective Equipment
Keywords: PPE; Multi-drug resistance organism; Cross-infection
MeSH Terms: conditions — COVID-19; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New PPE (Experimental): Use of Short sleeve gown and single pair of gloves
  Interventions: Other: New PPE
- Old PPE (Active Comparator): Use of Long sleeve gown and double pairs of gloves
  Interventions: Other: Old PPE

INTERVENTIONS:
Other: New PPE — The use of a new protocol of level 2 PPE which involves wearing a short-sleeve gown and a single pair of gloves
  Arms: New PPE
Other: Old PPE — The use of a standard protocol of level 2 PPE which involves wearing a long-sleeve gown and double pairs of gloves
  Arms: Old PPE

SUMMARY:
This study aims to improve the personal protective equipment (PPE) used while treating patients with COVID-19, to protect staff and avoid cross-infection of patients. Protecting staff from infection during the Covid pandemic is critical to maintaining health services. Mistakes in using protective equipment (PPE) are the commonest avoidable factor in staff becoming infected at work. Recently, intensive care doctors have also reported an increase in the spread of dangerous multi-resistant bacteria between patients, which appears likely to be transmitted between patients by Level 2 PPE worn by staff (specifically gown sleeves). This study therefore seeks to develop and test a new protocol to decrease cross-infection risks whilst using Level 2 PPE.

ELIGIBILITY:
Inclusion Criteria:

1. NHS staff and works in the Adult Intensive Care Unit, Neuro Intensive Care Unit or Cardio-thoracic Intensive Care Unit
2. Trained in the correct use of Level 2 PPE according to current guidance
3. Trained in ICU COVID19 Intubation and Proning protocols
4. Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. taking any medication which can cause photosensitivity reactions in the preceding 3 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants and simulated patients with contamination as assessed by ultraviolet light | immediately after simulations
  The primary outcome of this study is the proportion of participants and simulated patients who were contaminated with fluorescent powder as examined under a UV light, using a response of "YES" or "NO", when participants wore new (experimental) Level 2 PPE in comparison to the standard (control) Level 2 PPE

SECONDARY OUTCOMES:
Participants' perception of personal comfort and safety and safety of the patients as assessed through structured questionnaire | immediately before simulations and immediately after simulations
  We will measure the participants' perception of personal comfort and safety and the safety of the patient when wearing experimental versus control Level 2 PPE, during simulation tasks, using a 10 point Likert scale response to a structured questionnaire
changes in participants perception of personal comfort and safety and safety of patients as assessed through a semi-structured questionnaire | immediately before training, immediately after training and immediately after simulation
  We will measure changes in participants perception of their personal comfort and safety and the safety of patients when wearing each type of PPE using a semi-structured interview (a) before the PPE training, (b) after the PPE training, and (c) after the simulation training exercises.
The difference in the area of contamination between New and Standard PPE as analyzed through python script | immediately after simulations
  we will perform a quantitative analysis of the area of contamination of participants and simulated patients and assess the difference between when participants wore new (experimental) Level 2 PPE and the standard (control) Level 2 PPE, using pre-coded functions with python script.

CONTACTS AND LOCATIONS:
Overall Officials: Peter McCulloch, Principal Investigator — University of Oxford
Locations (1):
- Professor Peter McCulloch, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No